CLINICAL TRIAL: NCT02688062
Title: NeuroRegen Scaffold™ With Bone Marrow Mononuclear Cells Transplantation vs. Intradural Decompression and Adhesiolysis in Patients With Chronic Spinal Cord Injury
Brief Title: NeuroRegen Scaffold™ With Bone Marrow Mononuclear Cells Transplantation vs. Intradural Decompression and Adhesiolysis in SCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: First Hospitals affiliated to the China PLA General Hospital (Other Government)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-SDSCI/IGDB
Record Dates: First submitted 2016-02-06; First posted 2016-02-23 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroRegen Scaffold with BMMCs transplantation (Experimental)
  Interventions: Biological: NeuroRegen Scaffold with BMMCs transplantation
- Surgical intradural decompression and adhesiolysis (Experimental)
  Interventions: Procedure: Surgical intradural decompression and adhesiolysis

INTERVENTIONS:
Biological: NeuroRegen Scaffold with BMMCs transplantation — Patients with chronic SCI (ASIA grade A) will receive NeuroRegen Scaffold with bone marrow mononuclear cells (BMMCs) transplantation after localized scars cleared and after surgery patients will undergo a comprehensive rehabilitation, psychological and nutritional measures.
  Arms: NeuroRegen Scaffold with BMMCs transplantation
Procedure: Surgical intradural decompression and adhesiolysis — Patients with chronic SCI (ASIA grade A) will receive intradural decompression and adhesiolysis surgery and after surgery patients will undergo a comprehensive rehabilitation, psychological and nutritional measures.
  Arms: Surgical intradural decompression and adhesiolysis

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of NeuroRegen Scaffold with bone marrow mononuclear cells (BMMCs) on neurological recovery following chronic and complete spinal cord injury, compared to the treatment of surgical intradural decompression and adhesiolysis only.

ELIGIBILITY:
Inclusion Criteria:

1. Completely spinal cord injury at the thoracic level as assessed by magnetic resonance imaging (MRI) and electrophysiology.
2. ASIA Impairment Scale (AIS) grade A.
3. Male or female, 18-60 years old.
4. No significant further improvement after injury and rehabilitation.
5. Patients with normal peripheral nerve function and without muscle atrophy.
6. Cardiovascular, respiratory, liver, kidney functions and laboratory examinations are within normal ranges.
7. No brain disease or mental disorder.
8. Ability and willingness to regular visit to hospital and follow up during the protocol procedures.
9. Patients signed informed consent.

Exclusion Criteria:

1. A current diagnosis of any primary diseases affecting limb functions (e.g., traumatic brain injury, cerebral hemorrhage, cognitive disorders or other central nervous system diseases).
2. Patients without any rehabilitation train after injury.
3. Remarkable muscle atrophy or fibrosis.
4. Degeneration of peripheral nerve function.
5. Allergic constitution.
6. Participation in any immunomodulator therapy or experimental drug treatment within 60 days prior to study.
7. Suffering diabetes, autoimmune diseases, tumor or severe hypertension.
8. Patients with severe heart, lung, liver or renal dysfunction are unable to meet the surgery standards.
9. Severe bleeding tendency or abnormal coagulation function.
10. Inflammation or skin ulcers at the surgical site.
11. Lactating and pregnant woman.
12. Poor compliance, difficult to complete the study.
13. Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvements in ASIA (American Spinal Injury Association) Impairment Scale | 24 months
Improvements in Somatosensory Evoked Potentials (SSEP) | 24 months
Improvements in Motor Evoked Potentials (MEP) | 24 months

SECONDARY OUTCOMES:
Improvements in Independence Measures | 1, 3, 6, 12, 18 and 24 months
  Functional Independence Measure (FIM) will be assessed before and after surgery.
Magnetic Resonance Imaging (MRI) | 1, 3, 6, 12, 18 and 24 months
  The change of treated spinal cord injury will be assessed by Magnetic Resonance Imaging (MRI) before and after surgery.
Improvements in Urinary and Bowel Function | 1, 3, 6, 12, 18 and 24 months
  The ability to feel and control urination and bowel will be assessed based on bladder pressure monitory before and after surgery.
Safety and Tolerability assessed by Adverse Events | Up to 6 months
  Proportion of patients with postoperative infections and serious adverse events (SAEs) will be assessed by long term follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D., Principal Investigator — Chinese Academy of Sciences
Locations (1):
- First Affiliated Hospital of PLA General Hospital, Beijing, China